CLINICAL TRIAL: NCT01883986
Title: Palliative Care Interventions for Outpatients With Newly Diagnosed Lung Cancer
Brief Title: Supportive Care for Patients Newly Diagnosed With Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRI 12-141
Record Dates: First submitted 2013-06-18; First posted 2013-06-21 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-12

CONDITIONS: Lung Cancer
Keywords: palliative care
MeSH Terms: conditions — Lung Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): This is a 3 month nurse-led telephone based program integrating palliative care into usual oncologic care for patients diagnosed within 2 months of any type and stage of lung cancer.
  Interventions: Behavioral: Palliative Care
- Usual Care (No Intervention): Subjects randomized to usual care will receive medical oncology, radiation oncology, pulmonary, CT surgery as indicated by the type of cancer. At the completion of 3 months of usual care, subjects are invited to join the intervention arm.

INTERVENTIONS:
Behavioral: Palliative Care — Care delivered by a nurse including symptom assessment and management, patient education on lung cancer and treatment options , discussion and communication about preferences for care, psychosocial assessment including referrals to ancillary services such as social services and spiritual care as requested by the patient.
  Arms: Intervention

SUMMARY:
The aims of this project are to assess the feasibility of recruiting patients and delivering a nurse-led telephone based palliative care intervention for patients with newly diagnosed lung cancer and to assess if among patients with newly diagnosed lung cancer, the investigators can estimate the effect of a nurse-led telephone based palliative care intervention on quality-of-life, symptom burden and patient satisfaction.

DETAILED DESCRIPTION:
Patients meeting entry criteria will be randomized to the intervention arm, palliative care plus usual care or the usual care arm. Patients randomized to the intervention arm will receive usual oncologic care and phone calls from a nurse. Outcomes measures will be collected at baseline, and 3 months.

The study will be performed at the VA Puget Sound Health Care System. The investigators will recruit individuals (n=40) with lung cancer over 1 year. The primary objective is to test the feasibility and acceptability of the intervention, and recruitment of subjects. The investigators will estimate the effect of a nurse-led telephone based palliative care intervention to improve quality-of-life, symptom burden and patient satisfaction. In addition, using validated instruments, the investigators will assess the potential effect size of the intervention on quality of provider communication and on clinician knowledge of patient preferences for life sustaining therapies. The results of this pilot study will inform a future randomized clinical trial to test the efficacy of the intervention on a larger scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed at the Puget Sound Health Care System with a primary diagnosis of lung cancer,
* any cell type or stage,
* diagnosed within 8 weeks of study enrollment.
* Must have telephone access,
* ability of understand English and
* provide informed consent.

Exclusion Criteria:

* Patients not eligible to participate in the study include those who are inpatients prior to randomization,
* those who are under the care of palliative care or hospice at the time of randomization,
* those who have severe mental health disorders,
* those who are unable to speak directly with the nurse over the telephone,
* or those that have the inability to provide informed consent. Investigators will recruit individuals (n=40) with lung cancer over a 12 month period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn F. Reinke, PhD ARNP, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 41 outpatients with lung cancer of any stage or type at the Puget Sound Health Care System within two months of diagnosis between 3/6/2014 and 9/1/2015. We reviewed weekly tumor board lists and consults to oncology and pulmonary services to mail invitation letters to eligible patients and then follow up by telephone.
Pre-assignment Details: Forty-one subjects completed informed consent and forty subjects were randomized. The subject who was consented, but not randomized, became ineligible by enrolling in hospice care.
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 20 (Allocated to intervention arm) | 20 (Allocated to usual care arm)
Did Not Complete Study | 3 | 1 (Did not completed study)
Completed | 17 (Received allocated intervention) | 19 (Completed study)
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (6) | 64.9 (17.6) | 66.7 (13.1)
Gender [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 19 | 19 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 19 | 18 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Lung Total Outcome Index Score at 3 Months
Description: Patient Quality of Life including symptoms as measured by the FACT-L (Functional Assessment of Cancer Therapy-Lung Scale). The FACT-L outcome measure reported is the mean change in the TOI subscale (Total Outcome Index) of the instrument, computed as the differences between final and baseline visit scores. The TOI subscale range is 0-84 with a higher score indicating a better quality of life.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 20 | 20
units on a scale | 2.7 (9.5) | 4.7 (17.7)

2. Secondary Outcome: Change From Baseline in Patient Satisfaction of Care at 3 Months
Description: Patient satisfaction with care will be assessed by using the FAMCARE- Patient Survey 13 (full unabbreviated scale name). The FAMCARE is a 13 item, 5 point likert-scale validated questionnaire measuring patient satisfaction with cancer care and assessing interactions with health care providers, performance status and symptom burden. Only total scores are reported (no subscales). The total scores range from 13-65 with scores of 52 > indicating satisfaction with care. The higher the score the better the outcome (better satisfaction with care). In full randomized clinical trials, the estimated minimal important difference is 5 points from baseline to 12 weeks.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 20 | 20
units on a scale | .76 (9.6) | 1.02 (7.2)

3. Secondary Outcome: Change in Baseline Quality of Clinician Communication at 3 Months
Description: The quality of clinician end-of-life communication will be measured from the patient's perspective by the Quality of Communication Questionnaire (QOC).The QOC consists of 13 items divided into two subscales, six general communication items and seven end-of-life topics. We analyzed the six-item "general communication skills" scale, which scores range from 0-10. The higher the score the better the provider's communication is. We asked patients to answer the questions in reference to the provider who was primarily responsible for managing their lung cancer.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 20 | 20
units on a scale | -.18 (1.91) | .39 (1.42)

4. Secondary Outcome: Change From Baseline in Clinician Knowledge of Patient Preferences at 3 Months
Description: Clinician knowledge of patient preferences for life sustaining treatments will be assessed at baseline and at the study end point by asking 2 validated questions to both the clinician and the patient and determining the level of agreement between the responses.
Time Frame: Baseline and 3 months
Population: No data was collected due to poor provider response to surveys.
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Intervention | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No